CLINICAL TRIAL: NCT06827847
Title: Comparative Evaluation of Shade Matching Using a Digital Spectrophotometer in Monochromatic Versus Polychromatic Layering Techniques for Restoring Fractured Incisal Angles of Maxillary Incisors: a Randomized Controlled Trial
Brief Title: Comparative Evaluation of Shade Matching Using a Digital Spectrophotometer in Monochromatic Versus Polychromatic Layering Techniques for Restoring Fractured Incisal Angles of Maxillary Incisors - Invivo Study
Acronym: Shade Matching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Abdelaziz, Associate Professor - Conservative Dentistry - Faculty of Oral and Dental Medicine, Badr University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUC-IACUC-250119-127
Record Dates: First submitted 2025-01-25; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Class IV Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Universal shade dental composite technique (Active Comparator): patient received composite restoration done by received universal composite material
  Interventions: Procedure: Traditional polychromatic layering dental composite technique; Procedure: Contemporary monochromatic single shade dental composite technique

INTERVENTIONS:
Procedure: Traditional polychromatic layering dental composite technique — patient received composite restoration done by layering technique
Procedure: Contemporary monochromatic single shade dental composite technique — patient received composite restoration done by single shade composite

SUMMARY:
The color and appearance of a tooth is complex phenomenon which is related to many factors such as color stability, The Blending Effect, color Induction, color assimilation effect of resin composite materials which are all fall under the Term Chameleon Effect Which Enables Resin composite material to obtain a shade that bears a resemblance to the color of the surrounding tooth structure. The usage of different opacities and shades to match the tooth structure is very time consuming for both patient and clinician. However, any clinical effectiveness of any dental restorative procedures such as composite replacement is dependent on their physical, chemical and mechanical features which are highly proportional with oral environment and resin material properties.

DETAILED DESCRIPTION:
Resin Composite Material allow light scattering between Enamel and Dentin Which aid in Internal diffusion So That Resin Composite Material blend with the surroundings. The color alteration Also is directly proportional with light absorption to make it undetectable when blended with tooth structure A Significant disadvantage of resin composite restorations is highly susceptibility to staining and discoloration by the time and aging process in the oral environment. Color instability is one of the main reasons for replacing restorations, particularly in anterior teeth. There are several factors that affect the color stability of resin composite including intrinsic factors, namely the chemical make-up of the materials. Moreover, other extrinsic factors including smoking and poor oral hygiene, as well as the absorption of dyes from consuming foods and beverages in the oral cavity influence the color stability of resin composite restoration.

The color of any observed restoration is dedicated by light scattering between resin composite material and other substrates such as Tooth structure beneath restoration and other hard dental tissues. Natural teeth and resin composite material should share Three basic parameters Chroma , Hue and Value . Other Parameters effect on observation such as opacity, translucency, glossy surface should be put in consideration During resin based composite manufacturing.

This investigation sought to determine the effectiveness of three distinct approaches to shade matching when restoring class iv in dental maxillary incisors using universal Universal shade dental composite technique, traditional polychromatic layering dental composite technique, and contemporary monochromatic single shade dental composite technique.

ELIGIBILITY:
Inclusion Criteria:

* fractured incisal angles in vital maxillary permanent incisors
* aged 16 to 35
* exhibits good oral hygiene

Exclusion Criteria:

* individuals with nonvital or endodontically treated teeth
* active periodontal disease
* significant medical complications
* malocclusion
* parafunctional habits

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Shade matching | 1 day
  Shade selection will be evaluated using Vita Easyshade which is a hand-held digital spectro-photometer that consists of a hand piece connected to a base unit by a monocoil fiber optic cable assembly with a probe tip of about 5 mm in diameter, before and after putting esthetic restorations, then different resin composite shading systems will be used in this study

CONTACTS AND LOCATIONS:
Locations (1):
- Badr University in Cairo (BUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No